CLINICAL TRIAL: NCT01781312
Title: Proof-of-concept Study of Efficacy and Safety of Dietary Supplementation With Probiotics in IgAN Patients
Brief Title: Probiotics in IgA Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uppsala University Hospital (Other)
Collaborators: University Hospital, Linkoeping (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Hilde Kloster Smerud, Clinical Research Scientist, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SMR-2712; SMR-2712 (Other: Protocol writer)
Record Dates: First submitted 2013-01-16; First posted 2013-01-31 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ProTectis (Experimental)
  Interventions: Dietary Supplement: ProTectis
- Gastrus (Experimental)
  Interventions: Dietary Supplement: Gastrus

INTERVENTIONS:
Dietary Supplement: ProTectis
  Arms: ProTectis
Dietary Supplement: Gastrus
  Arms: Gastrus

SUMMARY:
Recent studies have shown an increased gastrointestinal reactivity and increased intestinal permeability in IgA nephropathy (IgAN). Probiotic supplementation is known to impact the gastrointestinal immune system possibly by improvement of both the immunologic and the non-immunologic intestinal barrier. Probiotic supplementation should thus theoretically have an effect on IgAN. In this study the investigators will study the efficacy and safety of Lactobacillus reuteri.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years
* Primary IgAN, verified by biopsy
* Albuminuria > 0.75 g/24 h (verified by at least four sample results within a two years period prior to inclusion)
* Serum creatinine less than 200 umol/L (verified by at least four sample results within a two years period prior to inclusion)
* Having signed informed consent form

Exclusion Criteria:

* Participation in another clinical intervention trial
* Patients with celiac disease
* Patients with secondary IgAN
* Creatinine clearance below 30 ml/min (mean of 3 measurements)
* Introduction of an ACE inhibitor or angiotensin II receptor blocker during the last three months prior to inclusion
* Patients treated with immunosuppressive or systemic corticosteroid drugs within the last twelve months
* Patients using probiotic products within the last three months (includes probiotic milk products)
* Known allergy or intolerance to any of the ingredients in the probiotic product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-07 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Change in albuminuria | Baseline and 3 months

SECONDARY OUTCOMES:
Change in renal function | Baseline and 3 months
Change in IgA/IgG immune complexes | Baseline and 3 months
Change in hematuria | Baseline and 3 months
Change in immunological markers in blood | Baseline and 3 months
Change in IBS (irritable bowel syndrome) symptoms | Baseline and 3 months

OTHER OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 months and 5 months

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - Linköping University Hospital, Linköping
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hosptial, Uppsala